CLINICAL TRIAL: NCT06015451
Title: Exercise Interventions in Patients With Postconcussion Symptoms and Posttraumatic Headache. A Randomized Controlled Trial.
Brief Title: Exercise in Postconcussion Symptoms and Posttraumatic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 468196
Record Dates: First submitted 2023-07-20; First posted 2023-08-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Brain Concussion; Post-Concussion Syndrome; Post-Traumatic Headache; Craniocerebral Trauma
Keywords: exercise intolerance; exercise; Thread mill test
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Post-Traumatic Headache; Craniocerebral Trauma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treadmill test after completion of intervention is performed by an assessor that is blinded for group membership.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow-up face-to face (Active Comparator): Home-based and in-house exercise, supervised both by telephone and face-to-face.
  Every week the first three weeks participants will exercise one session at the hospital, and the BCTT/BCCT will be performed every 3rd week, at the hospital in order to be able to shape the intervention.
  Interventions: Other: Sub-symptom threshold exercise
- Follow-up over the phone (Active Comparator): Home-based exercise only, supervised by telephone. The participants will exercise solely in the home setting and will be contacted by telephone, every week during the first three weeks, thereafter every third week. Based on the therapist's evaluation during these calls, the intervention is shaped.
  Interventions: Other: Sub-symptom threshold exercise

INTERVENTIONS:
Other: Sub-symptom threshold exercise — Aerob exercise at an intensity just below the intensity that provokes symptom exacerbation.

SUMMARY:
The goal of this clinical trial is to compare two models of delivery of guided exercise in patients with exercise intolerance after mild head injury.

The main question it aims to answer is:

• Is a program that includes elements of in-house exercise and follow-up sessions, and repeated treadmill testing, superior to a program with telephone-based follow-up only?

Participants will undergo a treadmill test to determine eligibility for the study, and to determine at what intensity level their symptoms worsen (symptom threshold). Thereafter they will exercise 15-20 minutes, 3-5 times per week at 80-90% of the heart rate that was found to be the symptom threshold. One group will receive face-to-face folllow-up and repeated testing, one group will receive telephone-based follow-up only .

Researchers will compare these two groups to see if closer follow-up is superior when it comes to recovery from exercise intolerance after 12 weeks of exercise.

DETAILED DESCRIPTION:
Patients with self-reported symptom exacerbation in relation to physical activity will be screened for inclusion with Buffalo Concussion Treadmill test (BCTT), an incremental treadmill exercise test according to a standard Balke protocol, to the first sign of symptom exacerbation or submaximal exertion. Heart rate and perceived exertion (Borg scale) are measured every minute. Patients who demonstrate symptom exacerbation according to predefined criteria will receive an individually tailored program for workouts with self-selected aerobic activites, of 15-20 minutes duration, 4-5 times per week at 85-90% (measured with HR monitor) of the HR at test termination, and they are randomised to either:

A. Every week the first three weeks, participants will exercise one individual session at the hospital, and the BCTT will be performed every 3rd week at the hospital to be able to shape the intervention.

B. The participants will only exercise at home, and will be contacted by telephone/video call, every week during the first three weeks, thereafter less often, up to every third week.

After 12 weeks, there will be a repeated BCTT, performed by a blinded assessor.

Patient reported outcomes are collected using electronic questionnaires before and after the intervention and 6 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Having sustained a minimal head injury or mild traumatic brain injury at least 2 weeks ago.
* At least one postconcussion symptoms, of at least moderate degree, occurring within the first week after the head injury.
* Intolerance for physical activity (self-reported and measured; including symptom exacerbation later on the test day).
* Capable of giving informed consent.

Exclusion Criteria:

* More than 2 years since last injury.
* The symptoms are better explained by other conditions.
* Severe communication problems, typically due to poor knowledge of Norwegian.
* Severe psychiatric, neurological, somatic, or substance abuse disorders that will make it problematic to function in a group and/or will complicate follow-up and outcome assessment.
* Safety concerns according to the study medical checklist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | 3 months
  Change in heart rate at test termination (the Buffalo Concussion Treadmill Test)

SECONDARY OUTCOMES:
Headache burden | 6 months
  Change in days of headache of at least moderate intensity
Change on self-selected area of function. | 6 months
  Change on the Patient-specific Function Scale (PSFS), the first 3 items, range 0-30, highest is worst.
Self-reported amount of physical activity | 6 months
  Change on the International Physical Activity Questionnaire (IPAQ), higher total values indicate more physical activity.
Quality of life after head injury (QOL) | 6 months
  Change on the Quality of life after brain injury - Overall Scale (QOLIBRI - OS). Six items rated on an ordinal scale, higher score indicate better QOL.
Depressive symptoms | 6 months
  Change on the Patient Health Questionnaire (PHQ-9). Nine items range 0-3, higher score indicates more severe depressive symptoms.
Anxiety | 6 months
  Change on the Generalized Anxiety Disorder Scale (GAD-7). Seven items range 0-3, higher score indicates more severe symptoms of anxiety.
Impact of headaches | 6 months
  Change on the Headache Impact Test (HIT)-6. Six items, Total score ranges from 36-78, higher score indicates higher impact.
Fatigue | 6 months
  Change on the Fatigue Severity Scale (FSS). Nina items, total score range 9-63, higher score indicates more severe fatigue.
Adherence to training | 6 months
  The Problematic Experience of Therapy scale (PETS). 12 questions with responses on a Likert scale. No total score.

CONTACTS AND LOCATIONS:
Overall Officials: Britt-Elin Lurud, MD, Study Director — Clinic of Rehabilitation, St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Clinic of Rehabilitation, Trondheim, Norway

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT06015451/Prot_SAP_000.pdf